CLINICAL TRIAL: NCT06186817
Title: Effectiveness of Manual Therapy Based on the Fascial Distortion Model on the Cervical Spine in Individuals With Temporomandibular Disorder
Brief Title: Effectiveness of the Fascial Distortion Model on the Cervical Spine in Individuals With Temporomandibular Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Karabuk University (Other)
Responsible Party: Principal Investigator, Harun Gençosmanoğlu, Principal Investigator, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/1359
Record Dates: First submitted 2023-12-17; First posted 2024-01-02 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-07

CONDITIONS: Temporomandibular Disorder; Temporomandibular Disorders; Temporomandibular Joint Disorders; Temporomandibular Joint Dysfunction Syndrome; Temporomandibular Joint Dysfunction; Manual Therapy; Core Stabilization Exercise Therapy
Keywords: Temporomandibular Disorders; Fascial Distortion Model; Core Stabilization Training; Head Posture; Neck Pain; Manual Therapy
MeSH Terms: conditions — Temporomandibular Joint Disorders; Temporomandibular Joint Dysfunction Syndrome; Neck Pain | interventions — Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Manual Therapy based Fascial Distortion Model (Active Comparator): All participants were given manual therapy based on the Fascial Distortion Model in addition to conventional therapy (Rocabado's 6x6 Exercises and Patient Education). Conventional therapy was implemented as a home program for 8 weeks, while Manual Therapy was conducted for forty-five minutes once a week in a clinical setting.
  Interventions: Procedure: Fascial Distortion Model; Procedure: Rocabado's 6x6 Exercises; Behavioral: Patient Education
- Core Stabilization Training (Active Comparator): All participants were given manual therapy based on the Core Stabilization Training in addition to conventional therapy (Rocabado's 6x6 Exercises and Patient Education). Conventional therapy was implemented as a home program for 8 weeks, while Core Stabilization Training was conducted for forty-five minutes once a week in a clinical setting.
  Interventions: Procedure: Rocabado's 6x6 Exercises; Behavioral: Patient Education; Procedure: Core Stabilization Training
- Control (No Intervention): No participant was given any therapy during the study.

INTERVENTIONS:
Procedure: Fascial Distortion Model — The following techniques were used on the cranial and cervical areas during therapy: Trigger band technique, herniated trigger point technique, continuum technique, folding technique, cylinder technique, and tectonic technique.
  Arms: Manual Therapy based Fascial Distortion Model
Procedure: Rocabado's 6x6 Exercises — Resting position of the tongue, rotational control of temporomandibular joint, rhythmic stabilization, axial extension of the neck, shoulder posture, and stabilized head flexion
  Arms: Core Stabilization Training; Manual Therapy based Fascial Distortion Model
Behavioral: Patient Education — Participants are instructed to perform some behaviors while avoiding others based on the etiology of temporomandibular disorders.
  Arms: Core Stabilization Training; Manual Therapy based Fascial Distortion Model
Procedure: Core Stabilization Training — Week 1st (1 x 10 reps): Supine deep cervical activation, supine deep lumbar activation, prone deep cervical activation, prone deep lumbar activation, supine combined deep cervical and lumbar activation, and prone combined deep cervical and lumbar activation; Week 2nd (1 x 10 reps): Arm openings, hundreds 1, one leg stretch 1, double leg stretch 1, shoulder bridge, breaststroke, leg pull prone prep 1; Week 3rd (1 x 10 reps): Arm openings, hundreds 2, one leg stretch 2, double leg stretch 2, shoulder bridge, breaststroke, leg pull prone prep 2; Week 4th (1 x 10 reps): Arm openings, hundreds 2, one leg stretch 2, double leg stretch 3, shoulder bridge, breaststroke, leg pull prone prep 2; Week 5th to 8th (with Resistance Band; 1 x 10 reps): Arm openings, shoulder bridge, swan dive, scapula isolations, plough, biceps curl, roll up, roll up with biceps, roll up with rowing, seated spine twist, swimming in kneeling, one leg kick in kneeling and diamond press in standing
  Other Names: Spinal Stabilization Training
  Arms: Core Stabilization Training

SUMMARY:
The goal of this randomized clinical trial is to investigate the effectiveness of Manual Therapy Based on the Fascial Distortion Model (FDM) on the cervical spine by comparing it with Core Stabilization Training (CST) or Control in individuals with temporomandibular disorders. The main questions it aims to answer are:

Is the effectiveness of the addition of FDM-based Manual Therapy to conventional therapy different from the addition of CST or control? Is the effectiveness of the addition of CST to conventional therapy different from the addition of FDM or control? All participants in the intervention groups will be given eight-week conventional therapy (Rocabado Exercises and Patient Education) in addition to FDM-based Manual Therapy or CST. Participants in the control group will not be given any therapy during the study.

Neck pain intensity, hand grip strength, head posture, cervical muscle performance, cervical range of motion (function), disability, and quality of life will be assessed.

DETAILED DESCRIPTION:
Interventions are needed to address neck pain intensity, hand grip strength, head posture, cervical muscle performance, cervical range of motion (function), disability, and quality of life in individuals with temporomandibular disorder (TMD). This study aims to examine the effectiveness of Fascial Distortion Model-based Manual Therapy compared to Core Stabilization Training or Control in individuals with TMD over an 8-week period. Individuals with TMD will be randomized into Group 1 (Fascial Distortion Model-based Manual Therapy, Rocabado Exercises, and Patient Education), Group 2 (Core Stabilization Training, Rocabado Exercises, and Patient Education), or Group 3 (Control). Rocabado Exercises and Patient Education will be implemented as a home program for 8 weeks, while Fascial Distortion Model-based Manual Therapy and Core Stabilization Training will be conducted once a week in a clinical setting. Neck pain intensity will be assessed using the Graded Chronic Pain Scale (Revised) and the Short-Form McGill Pain Questionnaire. Hand grip strength and head posture will be assessed using a hand dynamometer and lateral photography, respectively. The Functional Strength Testing of the Cervical Spine and cervical range of motions will be used to assess cervical muscle performance and function, respectively. Disability and quality of life will be evaluated using the Neck Disability Index and the Cognitive Exercise Therapy Approach-Biopsychosocial Questionnaire. All outcomes will be measured at baseline and end of the study, while neck pain intensity will also undergo intermediate assessments (2nd, 4th, and 6th weeks).

ELIGIBILITY:
Inclusion Criteria:

* Having a temporomandibular joint complaint that has persisted for three months
* Being diagnosed with temporomandibular disorder according to the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) Axis I
* Comprehension and interest in responding to assessment questions

Exclusion Criteria:

* Having a systemic condition (neurological, rheumatological, oncological, etc.) that could affect the temporomandibular joint and/or interfere with the evaluation
* History of any trauma that may have affected cranial, cervical, or facial region
* Having undergone any surgical intervention in cranial, cervical, or facial regions in the previous six months
* Receiving any surgical treatment, medical treatment, or physiotherapy for temporomandibular disorder in the last month
* Having received radiotherapy in the cranial or cervical region
* Pregnancy or breastfeeding
* Exercise for head posture for the last month

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2023-12-17 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2025-01-02 (Actual)

PRIMARY OUTCOMES:
Eye-Tragus-Horizontal Angle on lateral photography of head posture | From enrollment to the end of treatment at 8 weeks
  The angle between the line connecting the midpoint of the lateral corner of the eye to the tragus of ear and the horizontal line emerging from the tragus level. It refers to the cranial rotation angle
Pogonion-Tragus-C7 Angle on lateral photography of head posture | From enrollment to the end of treatment at 8 weeks
  The angle between the line connecting the pogonion (the most protruding point on the front of the mandible) to the tragus and the line connecting the tragus to the C7 vertebra
Tragus-C7-Horizontal Angle on lateral photography of head posture | From enrollment to the end of treatment at 8 weeks
  The angle between the line connecting the tragus to the C7 vertebra and the horizontal line emerging from the C7 vertebra level. It refers to the neck inclination angle
Tragus-C7-Shoulder Angle on lateral photography of head posture | From enrollment to the end of treatment at 8 weeks
  The angle between the line connecting the acromion to the C7 vertebra and the line connecting the C7 vertebra to the tragus. It refers to the sum of the tragus-C7-horizontal angle and the shoulder-C7-horizontal angle; Shoulder-C7-Horizontal Angle (5): The angle between the line connecting the acromion to the C7 vertebra and the horizontal line emerging from the C7 vertebra level. It refers to the angle of the shoulder.
Shoulder-C7-Horizontal Angle on lateral photography of head posture | From enrollment to the end of treatment at 8 weeks
  The angle between the line connecting the acromion to the C7 vertebra and the horizontal line emerging from the C7 vertebra level. It refers to the angle of the shoulder.
Disability based on Neck Disability Index | From enrollment to the end of treatment at 8 weeks
  Neck Disability Index. Minimum and maximum values are 0 and 5 points, respectively. Higher scores mean a worse outcome.
Quality of Life based on Cognitive Exercise Therapy Approach-Biopsychosocial Questionnaire | From enrollment to the end of treatment at 8 weeks
  Cognitive Exercise Therapy Approach-Biopsychosocial Questionnaire. Minimum and maximum values are 0 and 4 points, respectively. Higher scores mean a worse outcome.
Chronic neck pain intensity | Baseline, 2nd week, 4th week, 6th week and 8th week
  Graded Chronic Pain Scale (Revised). Scoring: Grade 1=mild, Grade 2=bothersome, Grade 3=high impact chronic pain. Higher scores mean a worse outcome.
Neck pain intensity at last seven days based on Short-Form McGill Pain Questionnaire | Baseline, 2nd week, 4th week, 6th week and 8th week
  Short-Form McGill Pain Questionnaire. Minimum and maximum values are 0 and 3 points, respectively. Higher scores mean a worse outcome.
Present neck pain intensity | Baseline, 2nd week, 4th week, 6th week and 8th week
  Visual Analog Scale. Minimum and maximum values are 0 and 10 cm, respectively. Higher scores mean a worse outcome.
Present neck pain intensity (ordinal) | Baseline, 2nd week, 4th week, 6th week and 8th week
  Present pain intensity scale of McGill Pain Questionnaire. Minimum and maximum values are 0 and 5 points, respectively. Higher scores mean a worse outcome.
Neck pain intensity at last seven days based on Numeric Pain Rating Scale | Baseline, 2nd week, 4th week, 6th week and 8th week
  Numeric Pain Rating Scale. Minimum and maximum values are 0 and 10 points, respectively. Higher scores mean a worse outcome.
Cervical active range of motion | From enrollment to the end of treatment at 8 weeks
  Dijital inclinometric measurements. Flexion, extension, right and left lateral flexions and right and left rotations.

SECONDARY OUTCOMES:
Hand grip strength | From enrollment to the end of treatment at 8 weeks
  An hand dynamometer will be used to measure grip strength. Two measurements will taken with a 30-second rest between each trial, and the average of the three measurements will be recorded.
Cervical muscle performance | From enrollment to the end of treatment at 8 weeks
  The Functional Strength Testing of the Cervical Spine was used to evaluate the cervical muscle performance. This is a test that functionally evaluates cervical muscle strength. Results of this test are assessed as functional, functionally fair, functionally poor, and nonfunctional. Six-to-eight repetitions for the flexion test and 20-25 s holding time for the other tests indicate that the test result is functional. Three-to-five repetitions for the flexion test and 10-19 s holding time for the other tests indicate that the test result is functionally fair. One-to-two repetitions for the flexion test and 1-9 s holding time for the other tests indicate that the test result is functionally poor. Zero repetition for the flexion test and 0 s holding time for the other tests indicate that the test result is nonfunctional. Each test was terminated at onset of pain, and the relevant value was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Harun Gençosmanoğlu, PT, MSc, Principal Investigator — Karabük University
Locations (2):
- Turkey (Türkiye) (2):
  - Hacettepe University, Ankara
  - Karabük University, Karabük

IPD SHARING:
Plan to Share IPD: No